CLINICAL TRIAL: NCT00107965
Title: A Multi-center, Randomized, Double-blind, Parallel-group, Vehicle-controlled Study to Determine the Safety of PEP005 0.0025%, 0.01% and 0.05% Gel With Two Treatment Schedules, Day 1 & 2 or Day 1 & 8 Applications to Actinic Keratoses
Brief Title: Study to Determine the Safety of Two Applications of PEP005 Topical Gel to Actinic Keratoses
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peplin (Industry)
Responsible Party: Janelle Katsamas, Peplin
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PEP005-001; 2005/145
Record Dates: First submitted 2005-04-11; First posted 2005-04-12 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Actinic Keratosis
Keywords: Actinic Keratosis; Solar Keratosis; AK; Sun spots; PEP005; Topical; Dermatology
MeSH Terms: conditions — Keratosis, Actinic; Melanosis | interventions — 3-ingenyl angelate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (8):
- 1 (Experimental)
  Interventions: Drug: PEP005
- 2 (Experimental)
  Interventions: Drug: PEP005
- 3 (Experimental)
  Interventions: Drug: PEP005
- 4 (Placebo Comparator)
  Interventions: Drug: PEP005
- 5 (Experimental)
  Interventions: Drug: PEP005
- 6 (Experimental)
  Interventions: Drug: PEP005
- 7 (Experimental)
  Interventions: Drug: PEP005
- 8 (Placebo Comparator)
  Interventions: Drug: PEP005

INTERVENTIONS:
Drug: PEP005 — 0.0025% PEP005 Topical Gel (Day 1,2 application)
  Arms: 1
Drug: PEP005 — 0.01% PEP005 Topical Gel (Day 1,2 application)
  Arms: 2
Drug: PEP005 — 0.05% PEP005 Topical Gel (Day 1,2 application)
  Arms: 3
Drug: PEP005 — Vehicle Gel (Day 1,2 application)
  Arms: 4
Drug: PEP005 — 0.0025% PEP005 Topical Gel (Day 1,8 application)
  Arms: 5
Drug: PEP005 — 0.01% PEP005 Topical Gel (Day 1,8 application)
  Arms: 6
Drug: PEP005 — 0.05% PEP005 Topical Gel (Day 1,8 application)
  Arms: 7
Drug: PEP005 — Vehicle Gel (Day 1,8 application)
  Arms: 8

SUMMARY:
The purpose of this study is to determine whether topical application of PEP005 is safe for the treatment of actinic keratoses.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients
* At least five individual AK lesions on the arms, shoulders, chest, face and/or scalp

Exclusion Criteria:

* A cosmetic or therapeutic procedure:

  * within 10 cm of the selected AK lesions during the 3 months prior to study entry or
  * anywhere during the 4 weeks prior to study entry or anticipated treatment during the study
* Treatment with 5-fluorouracil, imiquimod, diclofenac or photodynamic therapy:

  * of lesions located within 10 cm of the selected AK lesions during the 3 months prior to study entry or
  * anywhere during the 4 weeks prior to study entry or anticipated treatment during the study
* Use of acid-containing products, topical retinoids or light chemical peels within 10 cm of the selected AK lesions during the 3 months prior to study entry, or anticipated treatment in this same area during the study
* Treatment with immuno-modulators, cytotoxic drugs, or interferon/interferon inducers during the 4 weeks prior to study entry or anticipated treatment during the study
* Treatment with psoralen plus UVA or use of UVB therapy during the 6 months prior to study entry or anticipated treatment during the study
* Use of systemic retinoids during the 6 months prior to study entry or anticipated treatment during the study
* Anticipated excessive or prolonged exposure to ultraviolet light or use of topical salves, creams or ointments to the selected AK lesions during the study
* Females of childbearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-03; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
To determine the safety of PEP005 Topical Gel at 0.0025%, 0.01%, and 0.05% administered as two applications to patients with actinic keratosis (AKs) on the arms, shoulders, chest, face, and/or scalp | 85 days

SECONDARY OUTCOMES:
To evaluate the efficacy of PEP005 0.0025%, 0.01% and 0.05% Topical Gel in treating Actinic Keratoses | 85 days

CONTACTS AND LOCATIONS:
Overall Officials: Greg Siller, Principal Investigator
Locations (6):
- Australia (6):
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Siller Medical, Brisbane, Queensland
  - Skin and Cancer Foundation, Melbourne, Victoria
  - Monash Medical Centre, Melbourne, Victoria
  - Fremantle Dermatology, Fremantle, Western Australia
  - Private Dermaology Clinic, Fremantle, Western Australia